CLINICAL TRIAL: NCT02192320
Title: The Clinical Study of Atorvastatin and Dexamethasone on Treatment for Chronic Subdural Hematoma in the Patients With Coagulation Disorders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oriental Neurosurgery Evidence-Based-Study Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSDH2014
Record Dates: First submitted 2014-07-11; First posted 2014-07-16 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Subdural Hematoma
Keywords: Atorvastatin; Atorvastatin and Dexamethasone; Chronic Subdural Hematoma; conservative treatment
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Atorvastatin; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin and Dexamethasone (Experimental): Atorvastatin: 20 mg (every evening orally) for 5 weeks;
  Dexamethasone: 0.75mg Tid (1st-2nd week), 0.75mg Bid (3th week), 0.75mg Qd (4th week), 0.375mg Qd (5th week)
  Interventions: Drug: Atorvastatin and Dexamethasone
- Atorvastatin (Active Comparator): Atorvastatin: 20 mg (every evening orally) for 5 weeks
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 20 mg (every evening orally) for 5 weeks
  Arms: Atorvastatin
Drug: Atorvastatin and Dexamethasone — Atorvastatin: 20 mg (every evening orally) for 5 weeks;
  Dexamethasone:0.75mg Tid (1st-2nd week), 0.75mg Bid (3th week), 0.75mg Qd (4th week), 0.375mg Qd (5th week)
  Arms: Atorvastatin and Dexamethasone

SUMMARY:
To evaluate Efficacy and Safety of oral Atorvastatin and Dexamethasone on conservative treatment for Chronic Subdural Hematoma (CSDH) patients with Coagulation Disorders

DETAILED DESCRIPTION:
Study design: Two-arm,Evaluator-blinded study

Subjects: CSDH patients with Coagulation Disorders（Conservative treatment is adopted）

Sample size: 60 cases, 30 in Atorvastatin and Dexamethasone-treated group, 30 in Atorvastatin-treated group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and<90years old, both gender;
2. Long-term antiplatelet and anticoagulant drugs cause Coagulation Disorders;
3. CT scan reveals supratentorial, unilateral or bilateral chronic subdural hematoma (MRI scan is warranted if diagnosis is difficult);
4. The midline shift to less than 1 cm;
5. Attending physician makes a judgment that cerebral hernia would not occur and surgical operation might not be performed in a short time. Conservative treatment is adopted;
6. Patients have never undergo surgery on the hematoma;
7. Patient fully understood the nature of the study, and voluntarily participates and signs informed consent.

Exclusion Criteria:

1. Allergic to the statin and dexamethasone or its ingredients;
2. Hematoma caused by tumors, blood and other known comorbidities;
3. Abnormal liver function;
4. Uncontrolled hepatitis and other liver diseases, as well as suffering from other disease may interfere the study;
5. Patients have been on oral Statin treatment in the past four weeks;
6. Patients have been on oral Steroids treatment for a long time;
7. Diagnosed Diabetes patients with poorly controlled blood glucose
8. Participate in clinical trials in the past four weeks;
9. Pregnant or breastfeeding;
10. Failure of completing the trial by poor compliance;
11. For any reason, the researchers believe that the case is not suitable for inclusion.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Changes of hematoma volume | 2,5,12 weeks during treatment
  After 5 weeks' treatment, the hematoma will be assessed, then the therapy will be continued according to follow-up processes.Head CT to all the patients will be performed before the treatment, after the 2nd week and 5th week during treatment (at the end), at the 12th week during the follow-up.

SECONDARY OUTCOMES:
Outcome score (GOSE) in subjects | 2,5,12 weeks during treatment
Changes of peripheral blood for later tested SDF-1a, Treg, CXCR4 and related analysis | 2,5,12 weeks during treatment
Changes of neurological symptoms and signs | 2,5,12 weeks during treatment
Recurrence and prognosis of patient failure in those conservative treatment | 2,5,12 weeks during treatment
Outcome score (ADL-BI Scale) in subjects | 2,5,12 weeks during treatment

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality